CLINICAL TRIAL: NCT00483847
Title: TYGRIS - ROW: TYSABRI® Global Observational Program in Safety - Rest of World
Brief Title: TYGRIS - ROW: TYSABRI Global Observational Program in Safety - Rest of World
Acronym: TYGRIS - ROW
Status: Completed | Type: Observational
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: 101MS403
Record Dates: First submitted 2007-06-05; First posted 2007-06-07 (Estimated); Last update posted 2015-04-13 (Estimated); Status verified 2015-04

CONDITIONS: Multiple Sclerosis
Keywords: TYGRIS - Rest of World (ROW); TYSABRI; natalizumab; Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objective of this study is to determine the incidence and pattern of serious infections, malignancies, and other serious adverse events (SAEs) in participants with multiple sclerosis (MS) treated with TYSABRI (natalizumab).

DETAILED DESCRIPTION:
The TYSABRI Global Observational Program in Safety for Rest of World (TYGRIS - ROW)is a safety observational cohort program designed to obtain long-term safety data in multiple sclerosis (MS) participants treated with TYSABRI in a clinical practice setting in countries other than the United States and Canada.

The Prescribing Physician will collect participant information at routine clinic visits (using standard data collection tools) at approximately 6-month intervals for 5 years from the first TYSABRI infusion.

ELIGIBILITY:
Key Inclusion Criteria:

* All Multiple Sclerosis (MS) participants in Rest of World (ROW) who are prescribed and receiving TYSABRI in normal clinical practice at centers that are taking part in the study are eligible to participate in TYGRIS - ROW. Participants must have received at least 1 and not more than 3 infusions of TYSABRI.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Multiple Sclerosis (MS) participants treated with TYSABRI outside of North America
Sampling Method: Non-Probability Sample
Enrollment: 4296 (Actual)
Dates: Start 2006-09; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Number of participants with serious infections, malignancies, and other serious adverse events (SAEs) | 5 Years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- There are multiple sites throughout Europe in this clinical trial. Contact Advanced Medical Services (AMS)., Mannheim, Germany

REFERENCES:
- [Derived] Foley J, Carrillo-Infante C, Smith J, Evans K, Ho PR, Lee L, Kasliwal R, Stangel M, Vermersch P, Hutchinson M, Marinelli F, Smirnakis K; TYGRIS investigators. The 5-year Tysabri global observational program in safety (TYGRIS) study confirms the long-term safety profile of natalizumab treatment in multiple sclerosis. Mult Scler Relat Disord. 2020 Apr;39:101863. doi: 10.1016/j.msard.2019.101863. Epub 2019 Nov 21. PMID 31901758